CLINICAL TRIAL: NCT01655953
Title: Changes in Acid Base Status During High Salt Intake
Acronym: SL8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DLR German Aerospace Center (Other)
Collaborators: Charite University, Berlin, Germany (Other); University of Erlangen-Nürnberg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DLR Salty Life 8 Study
Record Dates: First submitted 2012-07-23; First posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Low Grade Metabolic Acidosis
MeSH Terms: interventions — potassium bicarbonate

ARMS (2):
- Campaign 1 (Experimental)
  Interventions: Dietary Supplement: High NaCl + KHCO3; Other: Control: high NaCl
- Campaign 2 (Experimental)
  Interventions: Dietary Supplement: High NaCl + KHCO3; Other: Control: high NaCl

INTERVENTIONS:
Dietary Supplement: High NaCl + KHCO3 — 7.7 mmol Na/kgBW/d + 90 mmol KHCO3
Other: Control: high NaCl — 7.7 mmol Na/kgBW/d

SUMMARY:
The study aimed to examine the effects of an alkalinisation of a NaCl (sodium chloride, salt)-rich diet on acid base status, bone metabolism, protein turnover and other influenced physiological systems. Due to increased urinary calcium excretion and bone resorption a high NaCl-intake is considered as a risk factor for osteoporosis. On the contrary an alkaline diet is known to have a beneficial influence on bone metabolism. Therefore the investigators hypothesized that an alkaline diet can reduce NaCl-induced bone resorption.

8 healthy male volunteers took part in a stationary study carried out in the metabolic ward of the German Aerospace Center. The study consisted of 2 campaigns, each lasting 16 days. Both campaigns were divided into 5 days of adaptation, 10 days of intervention and 1.5 days of stationary recovery. During the intervention period the volunteers diet was NaCl-rich (7.7 mmol Na/kg body weight/day) and supplemented in one campaign by 90 mmol potassium bicarbonate (KHCO3) in a randomized cross-over design. The other campaign served as control.

Bone metabolism was studied by bone formation markers in the fasting morning blood and 24h-urinary bone resorption markers. Acid base status was assessed by blood gas analyses in the fasted and the postprandial state as well as urinary markers. Protein turnover was studied with stable isotopes. Further physiological systems like energy metabolism and the cardiovascular system are also under investigation.

ELIGIBILITY:
Inclusion Criteria:

* healthy males
* 19 - 35 years
* 65 - 85kg
* 170 - 190 cm
* successfully completed psychological and medical screening

Exclusion Criteria:

* athletes
* smoking
* drug- or alcohol abuse
* hyperlipidemia
* renal diseases
* obesity
* anemia
* bone diseases
* diabetes
* rheumatism
* blood donation within three month prior to study start
* participation in another clinical investigation three month prior to study start

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2007-07; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change in daily urinary C- and N-terminal bone collagen telopeptides (mmol/d) | Daily for a duration of 16 days

SECONDARY OUTCOMES:
Serum concentration of bone specific alkaline phosphatase (microg/L) | Baseline, after 3, 6, 8, 10 days of intervention, 2 days after finishing the intervention
Daily Nitrogen balance (g/d) | Daily for a duration of 16 days
Free cortisol excretion in 24h urine (microg/d) | Baseline, after 3, 6, 10 days of intervention
Phenylalanine hydroxylation (micromol/min) | Baseline, end of intervention
Systolic blood pressure (bpm) | Daily for a duration of 16 days
24h urinary net acid excretion (mEq/d) | Baseline, end of intervention
Serum concentration of N-terminal propeptide Type I (mmol/L) | Baseline, after 3, 6, 8, 10 days of intervention, 2 days after finishing intervention
Free cortisone excretion in 24h urine (microg/d) | Baseline, after 3, 6, 10 days of intervention
Protein synthesis (micromol/min) | Baseline, end of intervention
Protein degradation (micromol/min) | Baseline, end of intervention
Diastolic blood pressure (bpm) | Daily for a duration of 16 days
Capillary pH | Baseline, after 3, 6, 8, 10 days of intervention, 2 days after finishing intervention
Capillary HCO3- Concentration (mmol/L) | Baseline, after 3, 6, 8, 10 days of intervention, 2 days after finishing intervention
Capillary Base excess (mmol/L) | Baseline, after 3, 6, 8, 10 days of intervention, 2 days after finishing intervention
Capillary pCO2 (mmHg) | Baseline, after 3, 6, 8, 10 days of intervention, 2 days after finishing intervention
Capillary pO2 (mmHg) | Baseline, after 3, 6, 8, 10 days of intervention, 2 days after finishing intervention

CONTACTS AND LOCATIONS:
Locations (1):
- German Aerospace Center (DLR), Cologne, Germany